CLINICAL TRIAL: NCT02903277
Title: National Observatory of Chronic Myeloid Leukemia Adolescent and Young Adults Treated With Tyrosine Kinase Inhibitors in First Intent
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-10
Record Dates: First submitted 2016-07-21; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The median age of onset of chronic myeloid leukemia (CML) in chronic phase PC is about 60 years. However CML affects all age groups including 18-25 year olds, called adult-young adolescents (AJA). In France, there is no record of CML and especially not for this particular population, only a European Register of CML in children up to 18 years has been set up under the coordination of Professor "Frederic Millot", pediatrics, CHU Poitiers. Malignancies diagnosed in this population usually have characteristics, evolution, therapeutic strategies with tyrosine kinase inhibitors (TKIs) are a real therapeutic revolution with an overall survival very significantly augmented but at present only a minority of patients may one day consider a final judgment of treatment. AJA are the most exposed patients to the complications, the socio-economic repercussions, professional and personal of a very long-term treatment. But there is little data in the literature concerning this population. Two studies show that diagnosis of CML presents with poor prognostic factors (high skoal), the observed responses are poorer compared to older patients but it is accompanied difference in survival in all cases with a decline of about 70 mois. However, these studies have focused solely on the patients included in the study receiving optimized treatment is not the standard treatment at the time. It is clearly demonstrated that the inclusion in a study brings a benefit to the patient. However, the majority of AJA are not included in a study. The investigators therefore want to describe the AYA population of CML in France and compare the evolution of patients included or not in a protocol. The investigators also want to investigate specific issues of the age of these patients as the reproductive desire. Indeed, while it does not seem to be any risk of teratogenicity for men treated with ITK, this risk is clearly established for women and requires specific supported. Another important point is that of the quality of life. The state of physical and mental health and his feelings, physical activity and its limitations and well-being was assessed by the SF-3612 questionnaire. The results of this analysis were compared with those already obtained for the general population (not representative of Italian adults with cancer sample) and adjusted for sex, age, geographic region, marital status and education level . There seems to be young people and women who express a feeling more pejorative. This does not only covers the frequency of side effects but also on physical activity and well-being. the affected population will be noted that that is particularly involved in the social, professional and in the development of his personal life. The impact of treatment on quality of life must be considered under penalty of seeing the difficulties of compliance. But several studies have demonstrated the negative impact of poor adherence in response to treatments .

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 30 years
* patients diagnosed with CML treated with TKI first line
* collecting their non-opposition

Exclusion Criteria:

* none

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients aged 18 to 30 years diagnosed with CML treated with a frontline ITK will be included in the observatory after collecting their non-opposition.
  In the retrospective part of the study, we will collect data from dead or lost to patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Collect clinical data of diagnosis of the AJA CML patients | Change from the inclusion at modification of treatment
  Describe the characteristics of the AJA CML patients (18-30 years) in terms of presentation at diagnosis, treatment choices, tolerance, adherence to therapeutic response, evolution and survival.
Treatment choices of the AJA CML patients | Change from the inclusion at modification of treatment
  Describe the characteristics of the AJA CML patients (18-30 years) in terms of presentation at diagnosis, treatment choices, tolerance, adherence to therapeutic response, evolution and survival.
Tolerance of treatments | Change from the inclusion at modification of treatment
  Describe the characteristics of the AJA CML patients (18-30 years) in terms of presentation at diagnosis, treatment choices, tolerance, adherence to therapeutic response, evolution and survival.
Adherence to therapeutic response | Change from the inclusion at modification of treatment
  Describe the characteristics of the AJA CML patients (18-30 years) in terms of presentation at diagnosis, treatment choices, tolerance, adherence to therapeutic response, evolution and survival.
Evolution of the disease | Change from the inclusion at modification of treatment
  Describe the characteristics of the AJA CML patients (18-30 years) in terms of presentation at diagnosis, treatment choices, tolerance, adherence to therapeutic response, evolution and survival.
Survival of the patient | Change from the inclusion at modification of treatment
  Describe the characteristics of the AJA CML patients (18-30 years) in terms of presentation at diagnosis, treatment choices, tolerance, adherence to therapeutic response, evolution and survival.